CLINICAL TRIAL: NCT03950752
Title: Effect of Consumption of Bagel Without Palm Oil on Postprandial Lipidemia in Healthy or With Mild-Moderate Hypertriglyceridemia Subjects. Postprandial, Randomized, Controlled, Crossover and Double-Blind Study (PALMFREE)
Brief Title: Effect of Consumption of Bagel Without Palm Oil on Postprandial Lipidemia
Acronym: PALMFREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Europastry S.A. (Unknown); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALMFREE
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Hyperlipemia
Keywords: postprandial; cardiovascular disease; saturated fatty acids; monounsaturated fatty acids; palm oil
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bagels with optimized composition in fatty acids (Experimental): Participants will consume three bagels with an optimized composition in fatty acids and without oil palm in only one day.
  Interventions: Combination Product: Optimized Bagel
- Bagels with conventional composition in fatty acids (Active Comparator): Participants will consume three bagels with a conventional composition in fatty acids in only one day.
  Interventions: Combination Product: Conventional Bagel

INTERVENTIONS:
Combination Product: Optimized Bagel — Participants will eat 132g of a bagel with an optimized composition in fatty acids in only one day, representing an ingestion of 556.5 kcal and 33g of total fat, of which 4.41g are saturated fatty acids, 24.27g are monounsaturated fatty acids, and 4.28g are polyunsaturated fatty acids.
  Arms: Bagels with optimized composition in fatty acids
Combination Product: Conventional Bagel — Participants will eat 132g of a bagel with a conventional composition in fatty acids in only one day, representing an ingestion of 589.0 kcal and 35.6g of total fat, of which 16.76g are saturated fatty acids, 13.00g are monounsaturated fatty acids, and 5.81g are polyunsaturated fatty acids
  Arms: Bagels with conventional composition in fatty acids

SUMMARY:
Postprandial lipemia produced by fat intake is a major risk factor for the development of cardiovascular diseases (CVD), the most important cause of disease and death in the Western world. Scientific evidence shows that the consumption of saturated fatty acids has a potential harmful effect on postprandial lipemia compared to the intake of monounsaturated fatty acids. The magnitude of postprandial lipemia is also determined by the health status of individuals, being altered in individuals with metabolic disorders associated with the development of CVD, such as hypertriglyceridemia.

Palm oil is widely used in bakery products because it is more economical compared to other fats and oils of other origin and for its stability properties that contribute to this type of food. This oil has a profile of fatty acids, rich in saturated fatty acids, mainly palmitic acid, which as mentioned above, is associated with health alterations. In addition, the investigators must add the environmental problems that are generated by the massive cultivation of the plant from which palm oil is extracted (oil palm Elaeis guineensis), including the loss of thousands of hectares of tropical forest and endangering to dozens of animal species from deforested areas.

The proliferation of all these arguments associated with the effect on the health and environment of the consumption of palm oil has given way to a paradigm shift in the use of palm oil in the food sector.

The hypothesis of the study is that consumption of bagels with a composition optimized in fatty acids, eliminating the content of palm oil and replacing it with high oleic sunflower oil and stearic acid completely hydrogenated without trans fatty acids, so that the same amount of fat is maintained, will decrease the postprandial lipemia, compared to the consumption of bagels with a more conventional composition in fatty acids, in healthy and / or with mild-moderate hypertriglyceridemia individuals.

The main objective of this study was to evaluate the effect of acute consumption of bagels without palm oil in its formulation and with an optimized fatty acid composition on postprandial lipemia measuring the evolution of plasma triglyceride levels in healthy and/or with mild-moderated hypertriglyceridemia individuals.

ELIGIBILITY:
Inclusion Criteria healthy population:

1. Men and women over 18 years of age.
2. Sign the informed consent.
3. Fasting serum triglyceride concentration < 150 mg/dL.

Exclusion Criteria healthy population:

1. Having diabetes (glucose ≥ 126 mg/dL).
2. BMI values <18 kg/m^2 o >25 kg/m^2.
3. Waist circumference > 150 cm.
4. Present dyslipidemia (LDL cholesterol > 189 mg/dL).
5. Present celiac disease or food allergies related to the study product.
6. Presenting anemia (hemoglobin ≤ 13 g/dL in men and ≤ 12 g/dL in women).
7. Being pregnant or intending to become pregnant.
8. Be in breastfeeding period.
9. Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
10. Follow a hypocaloric diet and/or pharmacological treatment for weight loss.

Inclusion Criteria mild-moderated hypertriglyceridemia population:

1. Men and women over 18 years of age.
2. Sign the informed consent.
3. Fasting serum triglyceride concentration ≥ 150 mg/dL.

Exclusion Criteria mild-moderated hypertriglyceridemia population:

1. Having diabetes (glucose ≥ 126 mg/dL).
2. Fasting serum triglyceride concentration > 880 mg/dL.
3. History of pancreatitis.
4. Serum LDL cholesterol levels > 189 mg/dL).
5. Present celiac disease or food allergies related to the study product.
6. Presenting anemia (hemoglobin ≤ 13 g/dL in men and ≤ 12 g/dL in women).
7. Being pregnant or intending to become pregnant.
8. Be in breastfeeding period.
9. Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
10. Follow a hypocaloric diet and/or pharmacological treatment for weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Postprandial triglycerides levels | Triglyceride levels in plasma will be determined before consuming bagels and after ingestion of bagels at 30 minutes, 1 hour, 2 hours, 4 hours and 6 hours at Visit 1 and Visit 2.
  Evolution of postprandial triglycerides levels in blood, assessed as area under the curve (AUC).
  Serum triglycerides levels will be measured by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).

SECONDARY OUTCOMES:
Changes in endothelial function | Endothelial function will be measured at 4 hours after the consumption of bagels at Visit 1 ad Visit 2.
  Measurement of the endothelial function using the Laser-Doppler technique.
Changes in blood pressure (measured in mmHg) | Blood pressure will be measured before consuming bagels and at 4 hours after the consumption of bagels at Visit 1 and Visit 2.
  Systolic and diastolic blood pressure (SBP and DBP) will be measured twice after 2-5 minutes of patient respite, seated, with one-minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Evolution of postprandial glucose and insulin levels | Glucose and insulin plasma levels will be determined before consuming bagels and at 30 minutes, 1 hour, 2 hours and 4 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evolution of postprandial glucose and insulin levels in blood. It will be measured as AUC.
  Serum glucose and insulin levels will be measured by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Evolution of postprandial non-esterified fatty acids, total cholesterol, LDL and HDL cholesterol blood levels. | Non-esterified fatty acids, total cholesterol, LDL and HDL cholesterol plasma levels will be determined before consuming bagels and at 1 hour, 2 hours, 4 hours and 6 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evolution of non-esterified fatty acids, total cholesterol, LDL and HDL cholesterol in blood after the consumption of bagels.
  Serum parameters will be measured by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Evolution of postprandial Apolipoprotein (Apo) B-48, Apo B100 and Apo A1 in blood. | Apo B48, Apo B100 and Apo A1 plasma levels will be determined before consuming bagels and at 4 hours and 6 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evolution of Apo B48, Apo B100 and Apo A1 in blood after the consumption of bagels.
  Apo B100 and Apo A1 in serum will be measured by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Apo B48 in serum will be measured by an ELISA kit.
Evolution of postprandial levels in blood of inflammation, thrombosis and oxidative stress markers in blood. | IL-6, E-selectin, ICAM, VCAM, PA-1, Thrombomodulin and ORAC plasma levels will be determined before consuming bagels and at 4 hours and 6 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evolution of the inflammation markers Interleukin 6 (IL-6), E-selectin, Intercellular adhesion molecule-1 (ICAM) and Vascular cellular adhesion molecule-1 (VCAM), the thrombosis markers Plasminogen activator 1 (PA-1) and Thrombomodulin, and the oxidative stress markers Oxygen Radical Absorbance Capacity (ORAC) and Malondialdehyde.
  Serum parameters will be measured by human ELISA kits.
Evolution of postprandial lipoprotein lipase activity in blood. | LPL activity levels in plasma wil be measurd before consuming bagels and at 4 hours and 6 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evolution of postprandial activity levels of lipoprotein lipase (LPL) in blood. It will measured by a fluorometric kit.
  Serum activity of LPL will be measured by an fluorometric kit.
Fatty acid composition of postprandial serum triglycerides levels in blood. | Fatty acid composition of serum triglycerides will be measured before consuming bagels and at 6 hours after the consumption of bagels at Visit 1 and Visit 2.
  Evaluation of fatty acid composition of serum triglycerides in blood. It will be measured by liquid chromatography coupled to mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — Centro Tecnológico de Nutrición y Salud (Eurecat_Reus). Reus, Tarragona, Spain.
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org